CLINICAL TRIAL: NCT00868387
Title: Effects of Macronutrient Relations on Body Weight, Body Composition, and Cardiovascular Risk Markers in Overweight Patients Attending a Telemedically Guided Weight Loss Program
Brief Title: Macronutrient Relations and Weight Loss in Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 003
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2013-12

CONDITIONS: Obesity
Keywords: weight reduction; low-carbohydrate; body fat; telemedicine; cardiovascular risk markers
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- energy-restricted, CHO-restricted diet (Experimental): Interventions: carbohydrate restriction of diet: 40% Frequency: daily Duration: 12 months
  Interventions: Other: energy-restricted, CHO-restricted diet
- energy-restricted, CHO-rich diet (Active Comparator): Comparator: carbohydrate content of diet: > 55% Frequency: daily Duration: 12 months
  Interventions: Other: energy-restricted, CHO-rich diet

INTERVENTIONS:
Other: energy-restricted, CHO-restricted diet — carbohydrate content of the diet < 40% Frequency: daily Duration: 12 months
  Arms: energy-restricted, CHO-restricted diet
Other: energy-restricted, CHO-rich diet — carbohydrate content of diet > 55% Frequency: daily Duration: 12 months
  Arms: energy-restricted, CHO-rich diet

SUMMARY:
The burden of overweight and obesity has dramatically increased during the last decades. High carbohydrate intake, particularly refined carbohydrates, probably increase the risk of obesity, type 2 diabetes, and metabolic syndrome. There is evidence that energy-restricted low-carbohydrate diets show greater weight loss and better improvement of cardiovascular risk markers compared to energy-restricted low-fat diets. Beside macronutrient relations, efficacy of weight loss programs depends on care and control. The investigators aim to investigate whether or not a carbohydrate-restricted telemedically guided weight loss program results in a more pronounced weight loss and influences metabolic risk markers more beneficial than a fat-restricted diet.

DETAILED DESCRIPTION:
see brief summary.

ELIGIBILITY:
Inclusion Criteria:

* age 18-70 years
* body mass index > 27 kg/m2

Exclusion Criteria:

* history of cardiovascular symptomatology
* cholelithiasis
* urolithiasis
* insulin dependent diabetes
* pacemaker implantation
* pregnancy
* lactation
* vegetarianism

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2005-11; Primary Completion 2006-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
body weight | 12 months

SECONDARY OUTCOMES:
waist circumference | 12 months
blood pressure | 12 months
blood lipids | 12 months
parameters of glucose metabolism | 12 months
fat mass | baseline, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Heinrich Koertke, PhD, Principal Investigator — Heart Center NRW
Locations (1):
- Heart Center North Rhine-Westfalia, Bad Oeynhausen, North Rhine-Westfalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Frisch S, Zittermann A, Berthold HK, Gotting C, Kuhn J, Kleesiek K, Stehle P, Kortke H. A randomized controlled trial on the efficacy of carbohydrate-reduced or fat-reduced diets in patients attending a telemedically guided weight loss program. Cardiovasc Diabetol. 2009 Jul 18;8:36. doi: 10.1186/1475-2840-8-36. PMID 19615091